CLINICAL TRIAL: NCT03808428
Title: CUHK Jockey Club Tech-Based Stroke Rehabilitation Programme for Elderly Centre - Interactive Exoskeleton Ankle Robot
Brief Title: CUHK Jockey Club HOPE 4 Care Programme - Ankle Robot
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chinese University of Hong Kong (Other)
Collaborators: The Hong Kong Jockey Club Charities Trust (Other)
Responsible Party: Principal Investigator, Raymond KY Tong, Professor and Chairman, Chinese University of Hong Kong
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2018.493
Record Dates: First submitted 2018-12-20; First posted 2019-01-17 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: Stroke
MeSH Terms: conditions — Stroke

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Ankle Group (Experimental): Integrated with force and motion sensors to identify gait phase and classify user walking intention using machine learning control algorithm.
  Interventions: Device: Ankle Group

INTERVENTIONS:
Device: Ankle Group — Provide sensory feedback to help subjects relearn how to walk in correct gait pattern.

SUMMARY:
The Hong Kong Jockey Club Charities Trust has supported CUHK to launch a three-year project 'CUHK Jockey Club HOPE4Care Programme' to implement four evidence-based advanced rehabilitation technologies in 40 local elderly day care centres and rehabilitation centres, to benefit the community. The Exoskeleton Ankle Robot is a robot-assisted Ankle-Foot-Orthosis to facilitate gait training of person after stroke with drop foot.

ELIGIBILITY:
Inclusion Criteria:

* have the ability to walk on the ground independently or with one personal assistance with or without walking aids
* able to understand simple commends

Exclusion Criteria:

* have other neurological, neuromuscular, and orthopedic diseases
* uncontrolled cardiovascular or respiratory disorders
* moderate to severe contractures in the lower extremities

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2019-02-01 (Estimated); Primary Completion 2021-12-31 (Estimated); Study Completion 2021-12-31 (Estimated)

PRIMARY OUTCOMES:
Fugl-Meyer Assessment Lower Extremity (FMA-LE) | 3-month follow-up

SECONDARY OUTCOMES:
Functional Ambulation Classification (FAC) | 3-month follow-up
Modified Ashworth Scale (MAS) | 3-month follow-up
Berg Balance Scale (BBS) | 3-month follow-up
Timed 10-Meter Walk Test (10MWT) | 3-month follow-up
6 Minute Walk Test (6MWT) | 3-month follow-up

CONTACTS AND LOCATIONS:
Overall Officials: Raymond Tong, PhD, Principal Investigator — Department of Biomedical Engineering, CUHK
Locations (1):
- Department of Biomedical Engineering, The Chinese University of Hong Kong, Hong Kong, Hong Kong

IPD SHARING:
Plan to Share IPD: No